### 1. Study Title

Association of the PaO□/PaCO□ Ratio With ICU Mortality Independent of Oxygen Saturation and Mean Arterial Pressure: A MIMIC-II Retrospective Cohort Study Acronym: RATIO-MIMIC

### 2. Study Objectives

### **Primary Objective:**

• To determine whether the PaO□/PaCO□ ratio is independently associated with ICU mortality in critically ill adults, adjusting for oxygen saturation (SpO□) and mean arterial pressure (MAP).

### **Secondary Objectives:**

- To explore the relationship between PaO□/PaCO□ ratio categories (e.g., tertiles
  or quartiles) and ICU length of stay.
- To perform subgroup analyses by mechanical ventilation status, age, or primary ICU diagnosis.

## 3. Study Design

• Type: Observational

Design: Retrospective cohort study

Population: Adult ICU patients (≥18 years) in MIMIC-II database

- **Sampling Method:** Retrospective census of all eligible patients meeting inclusion/exclusion criteria
- **Cohorts/Groups:** Single cohort; exposure analyzed as continuous and categorical (quartiles or tertiles)
- **Time Frame:** ICU admissions from 2001–2008 (MIMIC-II database)

# 4. Study Population

- Inclusion Criteria:
  - 1. Adult patients (≥18 years) at ICU admission
  - 2. First (index) ICU admission during hospitalization

 At least one arterial blood gas measurement with PaO□ and PaCO□ 4. Available SpO□ and MAP during ICU stay 5. Documented ICU discharge status **Exclusion Criteria:** 1. Age <18 years 2. Missing or non-numeric PaO□ or PaCO□ values 3. Missing ICU outcome data 4. Physiologically implausible ABG values 5. ECMO during ABG measurement (if identifiable) 6. No SpO□ or MAP measurements during ICU stay 7. Repeat ICU admissions beyond index stay 8. DNR/comfort-care orders prior to ABG measurement (optional for sensitivity analyses) 5. Data Collection and Variables **Exposure Variable:** PaO□/PaCO□ ratio (calculated from ABG measurements) Outcome Variable: ICU mortality (yes/no) Covariates for Adjustment: Oxygen saturation (SpO□) Mean arterial pressure (MAP) Age, sex, ICU type (medical/surgical), comorbidities (if available)

**Time Points:** First ABG per ICU stay (primary), or median/peak ABG values for

## 6. Statistical Analysis Plan (SAP)

sensitivity analysis

#### **6.1 Descriptive Analysis**

Continuous variables: mean ± SD or median (IQR)

Mechanical ventilation status

- Categorical variables: counts and percentages
- Compare baseline characteristics across PaO□/PaCO□ quartiles using ANOVA/Kruskal-Wallis for continuous variables and chi-square/Fisher's exact test for categorical variables

### **6.2 Primary Analysis**

- Model: Multivariable logistic regression
- **Dependent Variable:** ICU mortality (binary)
- Independent Variable: PaO□/PaCO□ ratio (continuous or categorical)
- Covariates: SpO□, MAP, age, sex, ICU type, comorbidities
- Effect Measures: Adjusted odds ratios (ORs) with 95% confidence intervals
- Assessment of Independence: Evaluate whether PaO□/PaCO□ remains statistically significant after adjustment

## 6.3 Secondary Analyses

- Subgroup Analyses: Mechanical ventilation status, age categories, ICU type
- Sensitivity Analyses:
  - Excluding extreme ABG values
  - Excluding DNR/comfort-care patients
  - Using alternative PaO□/PaCO□ calculation methods (first ABG vs. median ABG)
- Time-to-event Analysis (Optional): Cox proportional hazards for ICU length of stay, treating death as event

#### 6.4 Missing Data Handling

- Exclude patients missing primary exposure or outcome
- For covariates (SpO□, MAP, comorbidities):
  - If <5% missing: complete-case analysis</li>
  - If >5% missing: consider multiple imputation

#### 6.5 Statistical Software

- R (version ≥4.0) or STATA (version ≥16)
- Two-sided p-value < 0.05 considered statistically significant

### 7. Ethical Considerations

- Secondary analysis of de-identified public data (MIMIC-II)
- No new patient consent required
- Approved by MIT and Beth Israel Deaconess Medical Center Institutional Review Boards for public data use

# 8. Reporting

- Follow **STROBE guidelines** for observational studies
- Present baseline tables, regression results, and flowchart of included/excluded patients
- Include sensitivity and subgroup analyses
- Report odds ratios, 95% CI, and p-values